CLINICAL TRIAL: NCT06143332
Title: Domain-specific Aerobic Exercise Training in Coronary Artery Disease
Acronym: DOSE-EX-CAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Daniel Keir, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 123930
Record Dates: First submitted 2023-11-08; First posted 2023-11-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Moderate-intensity continuous training (Experimental): ~50 min of constant-power output cycling, 3 x per week at 85% of gas exchange threshold
  Interventions: Other: Aerobic exercise training
- Heavy-intensity continuous training (Experimental): 30 min of constant-power output cycling, 3 x per week at 70% of the difference between gas exchange threshold and respiratory compensation point
  Interventions: Other: Aerobic exercise training
- High (severe)-intensity interval training (Experimental): intervals; 4 x 4 min on - 3 min off at 115% of respiratory compensation point (work) and 50-70% gas exchange threshold (recovery)
  Interventions: Other: Aerobic exercise training

INTERVENTIONS:
Other: Aerobic exercise training — Aerobic exercise training on a cycle ergometer

SUMMARY:
Exercise training in cardiac rehabilitation (rehab) is a key part of managing a patient with heart disease. It has been shown that cardiac patients who increase their aerobic ("cardio") fitness by exercise training live longer, have better quality of life, and stay out of hospitals more than patients who do not improve their aerobic fitness. The more a patient improves their aerobic fitness the greater the benefit. But it has been shown that more than half of patients do not improve their aerobic fitness even after participating in cardiac rehab. This may be related to how hard patients are asked to train (their training "intensity"). The way intensity is chosen in current programs is commonly based on a "one-size fits all" method that may not consider that different patients have different abilities. There are more personalized methods to determine training intensity that exist, but these have never been used in cardiac rehab. One method divides intensity into three zones (zone 1 = moderate intensity; zone 2 = heavy intensity; zone 3 = very high intensity) that are based on when an individuals' biological responses to exercise change. The purpose of this study is to see if this approach gives better results in terms of changes in aerobic fitness and if training in the different zones makes a difference. Three groups of patients will be asked to train for 3 months in one of the three intensity zones. Aerobic fitness before and after exercise training will be compared to see which intensity zone results in the largest change.

DETAILED DESCRIPTION:
105 patients with coronary artery disease will randomized at a ratio of 1:1:1 to three months of personalized domain-based and work-matched training in the: 1) moderate-; 2) heavy-; and 3) severe-intensity domains. Age and sex-balance between groups will be achieved by stratified-block randomization

After randomization, the protocol is split in two. The "Testing" portion includes physiological, health, and anthropometric assessments acquired at baseline (i.e., week 0) and at weeks 7 and 14. The "Training" portion includes aerobic exercise training 3x per week on a cycle ergometer

Testing

Testing at weeks 0, 7, and 14 will be identical and completed over two days (Days 1 and 2).

On Day 1, blood will be drawn and analysed for resting plasma glucose, cholesterol, and lipid profiles. Next, participants will perform a "step-ramp-step" test that includes in series: a 6-min constant work rate bout at a low-intensity exercise (i.e., ~25 W) followed by a symptom-limited ramp-incremental test (~5-15 W·min-1); and, after 30 min of recovery, a 12-min constant-work rate bout of heavy-intensity exercise (i.e., above gas exchange threshold [GET] but below the respiratory compensation point [RCP], ~40% of peak power output). This protocol will provide measures of cardiorespiratory fitness (V̇O2peak, GET, RCP) and be used to identify and establish the work rate ranges associated with the moderate, heavy, and severe-intensity domains. Throughout the exercise protocol, participants will wear a 12-lead ECG and facemask from which respired gas fractions, flows, and volumes will be measured. Week 7 tests will be used to adjust training intensity.

Day 2 experiments will run 48-96 hours later. First, participants' body composition will be measured by Dual X-ray Absorptiometry. Next, participants will perform a step-incremental cycle test at 3 individual-specific work rates within each of the moderate-, heavy-, and severe-intensity domains. After a 4 min 10 W baseline, participants will complete 10 min of constant-work rate exercise at 85%GET (i.e., moderate), then 10 min of constant-work rate at 70% of the difference between GET and RCP (i.e., heavy), and then cycle for as long as they can at 115%RCP (i.e., severe; ~4-6 minutes). At select time points during the protocol, arterialized-venous blood will be sampled from a heated dorsal hand vein and immediately analyzed for blood gas and metabolite concentration using a blood gas analyzer. After each blood draw, participants' cardiac output (Q̇) will be measured non-invasively by open-circuit acetylene breathing. Following exercise, participants will be rested supine in a reclining chair and undergo carbon monoxide rebreathing to measure hemoglobin mass and calculate intravascular volumes.

Training

Total training duration is 12 weeks (weeks 1-6 and 8-13). All aerobic exercise training will be conducted at Western University. Gas exchange measurements obtained from the "Testing" Day 1 will be used to identify each patients' target training work rate(s). Exercise prescription for the 3 groups will be work-matched (i.e., equal in kJ) relative to moderate-intensity training and prescribed as follows: i) moderate (constant work rate for 50 min at 85%GET; MOD); ii) heavy (constant work rate for 25-35 min at ∆70; HVY); and iii) severe (intervals; 4 x 4 min on at 115% RCP - 3 min off at 50-70%GET; HIIT). After the training target is established, patients will train 3x per week on cycle ergometer in groups as large as 5.

Analyses

An ANCOVA with sex and baseline fitness as covariates will be used to compare post-training outcome variables of the RCT. The primary outcome measure is V̇O2peak; secondary outcomes measures include V̇O2 at GET and RCP; and tertiary outcome measures include: fasting blood lipids and glucose, adiposity, hematological variables, and submaximal and maximal alveolar and deadspace ventilation, Q̇, stroke volume, and a-vO2diff. Initial primary analysis will be according to randomization, regardless of adherence, for those who complete post-testing (intent-to-treat). However, to assess physiological effects of training intensities, a per-protocol analysis will be used in those who meet training adherence criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CAD who do not have any identified left ventricular dysfunction (i.e., left ventricular ejection fraction [LVEF] <50%) and who: were discharged from the hospital following admission for acute coronary syndrome (i.e., ST-elevation or non ST-elevation myocardial infarction, addressed with PCI or CABG, as documented by their attending physician; referred to St. Joseph's CRSP Program; completed a CPET at the St. Joseph's CRSP Program (as routine screening for cardiac rehabilitation) and have been cleared to exercise in a structured format (i.e., do not exhibit any contraindications to maximal exercise); without: respiratory or musculoskeletal issues that would prohibit them from cycling exercise.

Exclusion Criteria:

* Those who have: diagnosed heart failure, severe aortic stenosis, congenital coronary abnormality, 2-3° atrioventricular block, major arrhythmias such as atrial fibrillation (including paroxysmal), or are scheduled to undergo PCI or CABG surgery within 2 months following hospital discharge; are using insulin for diabetes; diagnosed with respiratory disease; or musculoskeletal issues that prohibit cycling exercise; and/or are unable to provide informed consent..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | baseline (week 0) and week 14
  Post-training peak oxygen uptake achieved during a symptom-limited incremental exercise test to task failure

SECONDARY OUTCOMES:
Positive responders | week 14
  The frequency of "positive" responders to exercise training in each exercise intensity domain-specific training group will be quantified and compared. Responsiveness will be determined by previously established CAD-specific minimal reliable changes for peak oxygen uptake
Gas exchange threshold | baseline (week 0) and week 14
  Post-training power output associated with the gas exchange threshold.
Respiratory compensation point | baseline (week 0) and week 14
  Post-training power output associated with the respiratory compensation point.

OTHER OUTCOMES:
Cardiac output | baseline (week 0) and week 14
  Post-training submaximal and maximal cardiac output measured by open-circuit acetylene breathing.
Stroke volume | baseline (week 0) and week 14
  Post-training submaximal and maximal stroke volume.
Arterio-venous oxygen difference | baseline (week 0) and week 14
  Post-training submaximal and maximal arterio-venous oxygen difference.
Hemoglobin mass | baseline (week 0) and week 14
  Post-training hemoglobin mass measured by CO rebreathing.
Fasting blood lipids | baseline (week 0) and week 14
  Post-training LDL, HDL, and total cholesterol and triglycerides
Body fat percentage | baseline (week 0) and week 14
  Post-training body fat percentage measured by dual x-ray absorptiometry.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No